CLINICAL TRIAL: NCT04093232
Title: Alterations in Knee Synovial Fluid Biomarkers and Volume Following Hymovis Injections Using a Pneumatic Assistive Compression Device and Ultrasound Guided Arthrocentesis: Correlation With Clinical Outcomes
Brief Title: Synovial Fluid Biomarkers Pre and Post Hymovis Knee Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Fidia Pharma USA Inc. (Industry)
Responsible Party: Principal Investigator, Richard Meehan, Professor of Medicine, National Jewish Health
Other Study IDs: HS 3179
Record Dates: First submitted 2019-09-10; First posted 2019-09-17 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid and peripheral blood samples will be cryopreserved for biomarkers of cartilage health and catabolic or anabolic protein measurements are to be correlated with clinical improvement post Hymovis injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Hymovis — All subjects will receive 2 ultrasound guided Hymovis injections and the goal of the study is to correlate responsiveness to subjects unique SF biomarker panel results before the first Hymovis injection and identify potential mechanism of action of those OA patients who receive the greatest benefit.

SUMMARY:
This NJH Investigator Initiated Study funded by Fidia will prospectively perform 2 ultrasound (US) guided knee aspirations in patients with knee osteoarthritis using a pneumatic compressive device (KneeTap ™) at baseline and at 3 months following 2 Hymovis® injections. Synovial fluid catabolic and anabolic proteins will be compared to those values in the peripheral blood and correlated with clinical outcome measurements at 3 ,6 and 12 months compared to baseline values; WOMAC, SF 36, visual analog pain scale, 6 minute walking distance and SF volumes quantitated by US.

DETAILED DESCRIPTION:
50 Subjects between 21-80 years with a BMI < 40 with mild to moderate knee osteoarthritis on x ray (KL grade II or III) will have a ultrasound guided arthrocentesis with an external pneumatic compression device (KneeTap) and if > 0.5 ml of synovial fluid is obtained they will received the first of 2 FDA approved Hymovis knee injections. A second ultrasound guided Hymovis intra-synovial space injection will be administered in one week with a repeat arthrocentesis in 3 months. Subjects will be compensated $ 50 for each of 4 of 5 study visits. Clinical outcome measures at study visits 1, 3 (3 months) 4 at (6 months) and 5 (12 months will include: VAS (Visual analog Global pain (1-10), SF -36 ,WOMAC questionnaires (Western Ontario and McMaster University Arthritis Index pain Scale), measured distance on 6 minute walking distance test and synovial fluid depth measured by ultrasound. The Synovial fluid biomarker panel will include values of over 45 separate cytokines,.chemokines and proteins from subjects pre vs post Hymovis injections and compared to values in the peripheral blood obtained simultaneously. SF biomarker analysis will be performed on cryopreserved samples using fluorescence multiplex bead based assays (Luminex) or by ELISA. All values as well as clinical outcome parameters will be entered into the REDCap system for statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate knee osteoarthritis on x ray
* age 21-80

Exclusion Criteria

* pregnant
* BMI > 40
* history of systemic immune disorders
* knee arthroplasty with replacement
* knee infection or surgery within 1 year
* glucocorticoid injection within 3 months inability to ambulate for 6 minutes without walking assistive devices
* unable to provide informed consent
* patients with a clinical contra-indication for an arthrocentesis or adverse reaction to prior intra-articular lidocaine or HA injections.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild to moderate(on x rays) symptomatic knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
WOMAC scores (Western Ontario and McMaster University Osteoarthritis Index) | Change from baselinescore values to those over 12 months
  Self reported numeric values: on pain, stiffness and 17 items of limitations on physical function scored as 0-5 (none, mild, moderate, severe or extreme)
SF 36 scores (Quality of Life Questionnaire) | Change from baseline score values to those over 12 months
  Self reported numeric values based upon multiple domains; assessment of over all health, 0-4, (excellent , very good, good, fair and poor) and score compared to the prior year, 0-4, (much better, somewhat better, about the same, somewhat worse, much worse) and 10 functional daily living activity questions with score 0-2, (not at all limited, limited a little, and limited a lot) and 4 questions on patients health compared to others expectations or worsen or excellent health and if they more easily become sick 0-4, (false, mostly false, don't know, mostly true or definitely true. Higher scores indicate worse health and disability.
VAS (Visual analogue scale) score for self reported pain | Change from baseline score values to those over 12 months
  Self Reported patient assessment of pain from 0 I(no pain) on the left to 10 worst pain ever. The paint selects their value on a continuous 10 cm line. A higher numeric number on a 0 -10 scale selected indicates more severe pain.
6 minute walking distance | Change in distance walked from baseline to that distance walked over 12 months
  The measured distance in meters walked during a 6 minute supervised walk on level ground.
Synovial fluid depth | Change in the depth of knee synovial fluid from baseline values to those at 12 months
  Ultrasound measurement in millimeters of the maximum SF depth during external pneumatic compression.

SECONDARY OUTCOMES:
Synovial fluid and peripheral blood biomarkers | Change in the baseline levels of biomarkers in pg/ml to the levels 3 months after the first of 2 Hymovis injections
  54 separate cytokines ,chemokines and proteins which can impact cartilage health will be measured in the synovial fluid by ELISA and Luminex multiplex platforms on cryopreserved samples to determine the levels of these catabolic inflammatory or anabolic proteins which may impact cartilage health.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Meehan, MD, Principal Investigator — Nnational Jewish health
Locations (1):
- national Jewish health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only de-identified SF cryopreserved samples may be made available to potential collaborators in the future.